CLINICAL TRIAL: NCT05420974
Title: Intraoperative Arthroscopic Near-infrared Fluorescence Imaging of the Vascular Perfusion of the Meniscus in Patients Treated With Meniscal Repair
Brief Title: NIR Arthroscopic Fluorescence Angiography of Menisci
Acronym: FLUORarth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Isala (Other)
Collaborators: Arthrex, Inc. (Industry); Diagnostic Green GmbH (Industry)
Responsible Party: Principal Investigator, Pieter B.A.A. van Driel, P.B.A.A. van Driel, MD, PhD, Isala
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL81068.07522
Record Dates: First submitted 2022-06-07; First posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Meniscus Rupture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NIR fluorescence (Experimental): The included patients will be subdivided in four equal subgroups in order to evaluate alteration of NIR fluorescence signal during arthroscopy in combination with a (temporary) tourniquet and irrigation pump system.
  Interventions: Procedure: NIR fluorescence imaging of the vascular perfusion of the meniscus using ICG

INTERVENTIONS:
Procedure: NIR fluorescence imaging of the vascular perfusion of the meniscus using ICG — NIR fluorescence imaging of vascular perfusion using the Arthrex NIR fluorescence scope and Indocyanin Green

SUMMARY:
This trial is an explorative single center, single-arm study to assess whether vascularization of the meniscus can be visualized intraoperatively using arthroscopic near-infrared (NIR) fluorescence using ICG during standard of care meniscal repair treatment.

DETAILED DESCRIPTION:
The meniscal healing process is based on two fundamental principles: a solid primary fixation, and a well-functioning biological process of cicatrization, where the presence of vascularization is thought to play a major role. Intra-operative near infrared fluorescence angiography using Indocyanine Green (ICG) is a widely used method for operative assessment of vascularization. Fluorescence guided detection of the vascularity surrounding a meniscal tear could be of great value to predict meniscal healing after repair.

This pilot study will explore the technical feasibility of intraoperative near-infrared fluorescence angiography of the meniscus in patients undergoing arthroscopic meniscal repair. Technical challenges for NIR fluorescence arthroscopy are the visibility of the vascular perfusion in microvessels in the dense meniscus, motion artifacts encountered with arthroscopy and wash in of ICG using a fluid irrigation system.

The included patients will be subdivided in four equal subgroups in order to evaluate alteration of NIR fluorescence signal during arthroscopy in combination with a tourniquet and/or irrigation pump system.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* Patients with on MRI confirmed Zone 1 meniscal tear
* Patients with a clinical indication for arthroscopic meniscal repair
* Before patient registration, written consent must be given according to ICH/GCP, national and local regulations.

Exclusion Criteria:

* Prior operative treatment of the ruptured meniscus
* Any condition that in the opinion of the investigator could potentially jeopardize the health status of the patient. In specific, these conditions concern smoking, diabetes and being overweight.
* Pregnancy
* allergy to iodine, shellfish or ICG;
* Psychological, familial sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
NIR fluorescence of the meniscus | Fluorescence imaging will be performed from 0-10 minutes after injection of ICG
  Detection of fluorescence in the meniscus (yes/no), determined intra-operatively during the arthroscopy procedure using NIR fluorescence imaging and ICG.

SECONDARY OUTCOMES:
T start | Fluorescence imaging will be performed from 0-10 minutes after injection of ICG
  Time between injection of ICG and initial detection of the fluorescence signal in the meniscus (T start).
I max | Fluorescence imaging will be performed from 0-10 minutes after injection of ICG
  Maximum fluorescence intensity (Imax) in the meniscus. Fluorescence intensity will be measured in arbitrary units as a mean of three different region of interests.
T max | 0-10 minutes
  Time to maximum intensity of the fluorescence signal
Baseline and End fluorescence intensity | Fluorescence imaging will be performed from 0-10 minutes after injection of ICG
  Baseline fluorescence intensity of the meniscus and the end fluorescence intensity in the meniscus
The ration between the maximum fluorescence intensity in the meniscus and the background fluorecence intensity. | Fluorescence imaging will be performed from 0-10 minutes after injection of ICG
  The fluorescence intensity is measured in arbitrary units as a mean of three region of interests.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Vahrmeijer AL, Hutteman M, van der Vorst JR, van de Velde CJ, Frangioni JV. Image-guided cancer surgery using near-infrared fluorescence. Nat Rev Clin Oncol. 2013 Sep;10(9):507-18. doi: 10.1038/nrclinonc.2013.123. Epub 2013 Jul 23. PMID 23881033
- [Result] Goncalves LN, van den Hoven P, van Schaik J, Leeuwenburgh L, Hendricks CHF, Verduijn PS, van der Bogt KEA, van Rijswijk CSP, Schepers A, Vahrmeijer AL, Hamming JF, van der Vorst JR. Perfusion Parameters in Near-Infrared Fluorescence Imaging with Indocyanine Green: A Systematic Review of the Literature. Life (Basel). 2021 May 11;11(5):433. doi: 10.3390/life11050433. PMID 34064948
- [Result] van Schie P, van der Lelij TJN, Gerritsen M, Meijer RPJ, van Arkel ERA, Fiocco M, Swen JA, Vahrmeijer AL, Hazelbag HM, Keereweer S, van Driel PBAA. Intra-operative assessment of the vascularisation of a cross section of the meniscus using near-infrared fluorescence imaging. Knee Surg Sports Traumatol Arthrosc. 2022 May;30(5):1629-1638. doi: 10.1007/s00167-021-06690-w. Epub 2021 Aug 4. PMID 34347140